CLINICAL TRIAL: NCT01323387
Title: Lumbar Degenerative Disc Disease Treated With
Brief Title: Lumbar Degenerative Disc Disease Treated With Anterior Tension Band System (ATB) With ALIF/FRA Spacer
Acronym: ATB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Synthes USA HQ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1255
Record Dates: First submitted 2011-03-23; First posted 2011-03-25 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Lumbar Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other): Interbody fusions with Anterior Plating
  Interventions: Device: Interbody Fusion

INTERVENTIONS:
Device: Interbody Fusion — allograft spacer + anterior plate
  Other Names: ATB; Anterior Tension Band

SUMMARY:
Multi-center, prospective nonrandomized study of treatment for 1 and 2 level degenerative disc disease between L2 and S1. Patients will be followed for a minimum of 2 years.

The primary objective of this study to measure fusion success in patients with lumbar degenerative disc disease using the ATB and ALIF/FRA Spacer. The Secondary objective is evaluation of the patient's quality of life, pain and function.

ELIGIBILITY:
Inclusion Criteria:

1. One or Two level (consecutive) degenerative disc disease between L2 and S1. Degenerative disc disease is defined as follows:

   Chronic pain (confirmed by patient exams and history) of discogenic origin, confirmed by radiographic evidence (e.g. MRI, discogram) two or more of the following:
   * Modic type 2 endplate changes on T2 weighted MRI
   * high intensity zone signal on T2 weighted MRI
   * positive discogram with negative controls
   * dark disc (diminished T2 weighted signal)
   * decreased disc height
2. Has experienced pain, functional deficit and/or neurological deficit for a minimum six month period of time prior to enrollment
3. Has failed to respond to non-operative treatment modalities for a minimum three month period of time prior to enrollment
4. Skeletally mature and at least 18 years of age
5. Signs the approved Informed Consent Document
6. Is available for long term follow-up and interval visits

Exclusion Criteria:

1. Has more than 2 levels to be instrumented
2. Has had a previous fusion attempt at the involved level(s)
3. Has had more than two previous open, lumbar spine surgical procedures at the involved level(s)
4. Currently implanted with anterior instrumentation at the involved level(s)
5. Patient would be classified as morbidly obese BMI > 35
6. Active localized or systemic infection
7. Presence of a disease entity or condition which significantly affects the possibility of bony fusion (e.g., osteoporosis, metastatic cancer, long-term use of steroids, etc.)
8. Has an immunosuppressive disorder
9. Pregnant or interested in becoming pregnant during the study.
10. Has a known sensitivity to device materials
11. Mentally incompetent or prisoner
12. Currently a participant in another study for the same indications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2004-04-01 (Actual); Primary Completion 2009-05-01 (Actual); Study Completion 2011-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirkham Wood, MD, Principal Investigator — Massachusetts General Hospital

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 178
Completed | 94
Not Completed | 84
Not completed — Withdrawal by Subject | 41
Not completed — Radiographic Data Unavailable | 1
Not completed — Revision | 14
Not completed — Protocol Violation | 12
Not completed — Randomized but Never Treated | 16

BASELINE CHARACTERISTICS:
Population: 178 subjects were enrolled in the study but 16 of these were never treated. A total of 162 subjects were both enrolled and treated.
  Of the 162 enrolled and treated subjects, 12 were excluded for protocol deviations. Therefore, the overall number of baseline participants was 150 subjects per protocol.
Arm/Group | Treatment
Number analyzed (Participants) | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 150
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 73
Region of Enrollment [Number; unit: participants]
  United States | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Successful Radiographic Fusion
Description: CT Scans and plain film x-rays will be evaluated. Demonstration of bridging trabecular bone through or external to the allograft spacer will be the measure of success.
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 94
Participants | 90

2. Secondary Outcome: Quality of Life Using the SF-12 Scale Physical Health Component Score (PCS). Number of Subjects Who Achieved 15% Improvement in PCS Compared to Baseline.
Description: Quality of Life using the SF-12 Scale Physical Health Component Score (PCS). The PCS is a measurement of health status with a range of 0-100. A higher score indicates less disability.
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Groups:
- Physical Health Composite Score (PCS): A self-reported quality of life assessment to measure a participant's interpretation of their physical well-being. A 15% improvement was considered a success.
Arm/Group | Physical Health Composite Score (PCS)
Number analyzed (Participants) | 92
Participants | 57

3. Secondary Outcome: Pain Scores on the Numeric Rating Scale (NRS)
Description: The Numeric Rating Scale (NRS) is a measurement of pain from a value of 0 (no pain) to a value of 10 (worst pain)
Time Frame: Baseline and 24 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 91
units on a scale
  NRS at Baseline | 8.0 (1.7)
  NRS at 24 Months | 4.6 (3.0)

4. Secondary Outcome: Oswestry Disability Index (ODI): Number of Subjects Who Achieved a 15% Improvement in ODI Compared to Baseline
Description: The outcome measure is the number of subjects who achieved a 15% improvement in ODI compared to baseline. The ODI is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain. ODI scores range from 0 to 100 with 0 equating to No Disability and 100 equating to the Maximum Disability Possible
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 92
Participants | 63

5. Secondary Outcome: Quality of Life Using SF-12 Scale (MCS): Number of Subjects Who Achieved 15% Improvement in MCS Compared to Baseline
Description: The outcome measure is the number of subjects who achieved a 15% improvement in MCS compared to baseline. The MCS (Mental Component Score) is a measurement of health status with a range of 0 to 100. A higher score indicates less disability.
Time Frame: Baseline and 24 Months
Measure: Count of Participants; unit: Participants
Groups:
- Physical Health Composite Score (MCS): A self-reported quality of life assessment to measure a participant's interpretation of their physical well-being. A 15% improvement was considered a success.
Arm/Group | Physical Health Composite Score (MCS)
Number analyzed (Participants) | 92
Participants | 42

6. Secondary Outcome: SF-12 Physical Composite Score (PCS) Summary
Description: The PCS (Physical Component Score) is a measurement of health status with a range of 0 to 100. A higher score indicates less disability.
Time Frame: Baseline and 24 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 92
Units on a scale
  PCS at Baseline | 29.4 (7.0)
  PCS at 24 Months | 38.9 (13.5)

7. Secondary Outcome: SF-12 Mental Composite Score (MCS) Summary
Description: The MCS (Mental Component Score) is a measurement of health status with a range of 0 to 100. A higher score indicates less disability.
Time Frame: Baseline and 24 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 92
Units on a scale
  MCS at Baseline | 38.2 (11.7)
  MCS at 24 Months | 45.6 (14.0)

8. Secondary Outcome: Oswestry Disability Index (ODI) Summary
Description: The Oswestry Disability Index (ODI) is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain. The scores can range from 0 to 100 with 0 equating to No Disability and 100 equating to the Maximum Disability Possible
Time Frame: Baseline and 24 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 92
Units on a scale
  ODI at Baseline | 53.3 (13.7)
  ODI at 24 Months | 31.8 (23.0)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 19/150
Other Adverse Events (participants affected / at risk) | 77/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=150)
Broken Components (Injury, poisoning and procedural complications) | 1 (1)
Device Slippage (Injury, poisoning and procedural complications) | 1 (1)
New Onset of Pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Pseudoarthrosis (Musculoskeletal and connective tissue disorders) | 10 (10)
Soft Tissue Damage (Musculoskeletal and connective tissue disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Vascular Injury (Vascular disorders) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Disc Fragment Dislodged (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=150)
New Onset of Pain (Nervous system disorders) | 38 (54)
Pseudoarthrosis (Musculoskeletal and connective tissue disorders) | 17 (17)
Vascular Injury (Vascular disorders) | 7 (7)
Numbness/Tingling Sensation (Nervous system disorders) | 5 (6)
Broken Components (Injury, poisoning and procedural complications) | 6 (7)
Infection (Infections and infestations) | 4 (4)
Neural Structure Injury (Nervous system disorders) | 4 (4)
Thrombosis/Thrombophlegitis (Vascular disorders) | 3 (3)
Adjacent Segment Degeneration (Musculoskeletal and connective tissue disorders) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Cysts Found in and around Spacer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Device Slippage (Product Issues) | 2 (2)
Disc Fragment Dislodged (Injury, poisoning and procedural complications) | 1 (1)
Edema (General disorders) | 1 (1)
Fracture of Vertebrae (Musculoskeletal and connective tissue disorders) | 2 (2)
Hematoma/Seroma (Blood and lymphatic system disorders) | 2 (2)
ileus (Gastrointestinal disorders) | 2 (2)
Insomnia (General disorders) | 2 (2)
Intestinal Blockage (Gastrointestinal disorders) | 1 (1)
Irregular Menstrual Cycle (Reproductive system and breast disorders) | 1 (1)
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Retrograde Ejaculation (Reproductive system and breast disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Soft Tissue Damage (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less